CLINICAL TRIAL: NCT01526655
Title: A Randomized Open Controlled Trial Comparing Robot Assisted Laparoscopic Hysterectomy and Abdominal Hysterectomy for Endometrial Cancer in a Fast Track Program
Brief Title: Robot Assisted Laparoscopic Hysterectomy vs. Abdominal Hysterectomy in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Preben Kjolhede, MD, professor, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROBOTHYST
Record Dates: First submitted 2012-01-28; First posted 2012-02-06 (Estimated); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-08

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Robot assisted laparoscopy; Abdominal hysterectomy; Fast track program
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominal total hysterectomy (Active Comparator): Standard extrafascial abdominal total hysterectomy through a low transverse abdominal wall incision
  Interventions: Procedure: Abdominal total hysterectomy
- Robot assisted laparoscopic hysterectomy (Active Comparator): Robot assisted laparoscopic total hysterectomy
  Interventions: Procedure: Robot assisted laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Abdominal total hysterectomy — Abdominal total hysterectomy through a low transverse abdominal wall incision
  Arms: Abdominal total hysterectomy
Procedure: Robot assisted laparoscopic hysterectomy — Robot assisted laparoscopic total hysterectomy
  Arms: Robot assisted laparoscopic hysterectomy

SUMMARY:
The purpose of the trial is to determine whether robot assisted laparoscopic hysterectomy compared with abdominal hysterectomy in a fast track program gives a faster recovery postoperatively, causes less tissue damage and less effects on the immunological system, and is health economically cost-effective.

DETAILED DESCRIPTION:
If detailed description is requested, please contact sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Scheduled to total hysterectomy + bilateral salpingooophorectomy (BSAE) and peritoneal lavage because of endometrial carcinoma, International federation of gynecology and obstetrics (FIGO) stage 1, grade 1 and 2, with diploid DNA profile (i.e. low risk profile).
* WHO (World Health Organisation) performance status ≤ 2.
* Proficiency in Swedish
* Accept to participate in the study and has signed written informed consent document.
* The operation should be considered possible to be perform laparoscopically and by laparotomy through a low transverse abdominal wall incision.

Exclusion Criteria:

* The operation is anticipated to comprise more than the hysterectomy + BSAE.
* A midline incision is planned for the laparotomy.
* Contraindications towards spinal anesthesia with intrathecally applied morphine.
* Physically disabled women who cannot be expected to be mobilized in accordance to the fast track program in a way similar to what is expected from not-physically disabled women.
* Mentally disabled women who cannot fill in the questionnaires or understand the consequences of participating in a trial.
* Severe psychiatric disease or on medication for psychiatric disease so that the physician consider participation in the trial inappropriate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, 58185 Linköping, Sweden; Evelyn Lundin, MD, Study Director — Department of Obstetrics and Gynecology, University Hospital, 58185 Linköping, Sweden; Ninnie Borendal Wodlin, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospital, 58185 Linköping, Sweden; Lena Nilsson, MD, PhD, Study Chair — Department of Anesthesiology, University Hospital, 58185 Linköping, Sweden; Jan Ernerudh, MD, PhD, Study Chair — Department of Clinical Immunology, University Hospital, 58185 Linköping, Sweden; Per Carlsson, PhD, Study Chair — Centre for Medical Technology Assessment, University Hospital, 58185 Linköping, Sweden
Locations (2):
- Sweden (2):
  - Department of Obstetrics and Gynecology, Ryhov Central Hospital, Jönköping, Jönköping County
  - Department of Obstetrics and Gynecology, University Hospital, Linköping, Östergötland County

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient withdrew consent prior to surgery in the control group (abdominal hysterectomy) and received the standard treatment.
Groups:
- Robotic Hysterectomy: Robot assisted laparoscopic total hysterectomy
- Abdominal Hysterectomy: Standard extrafascial abdominal total hysterectomy through a low transverse abdominal wall incision
Period: Overall Study
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 50 women with low-risk endometrial cancer scheduled for surgery between February 2012 and May 2016 were included.
Groups:
- Robotic Hysterectomy: Robot assisted laparoscopic total hysterectomy
  Robot assisted laparoscopic hysterectomy: Robot assisted laparoscopic total hysterectomy
- Abdominal Hysterectomy: Standard extrafascial abdominal total hysterectomy through a low transverse abdominal wall incision
  Abdominal total hysterectomy: Abdominal total hysterectomy through a low transverse abdominal wall incision
- Total: Total of all reporting groups
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 68 [38 to 83] | 67 [45 to 85] | 67 [38 to 85]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 25 | 25 | 50
Body mass index [Median (Full Range); unit: kg/m^2] | 28.2 [21.5 to 54.1] | 28.0 [19.4 to 37.8] | 28.1 [19.4 to 54.1]
Body mass index [Count of Participants; unit: Participants]
  BMI <25 | 7 | 8 | 15
  BMI 25-29.9 | 8 | 10 | 18
  BMI 30-35 | 6 | 5 | 11
  BMI > 35 | 4 | 2 | 6
Parity [Median (Full Range); unit: births] | 2 [0 to 5] | 2 [0 to 5] | 2 [0 to 5]
Smokers [Count of Participants; unit: Participants] | 4 | 0 | 4
Previous laparotomy [Count of Participants; unit: Participants] | 13 | 8 | 21
Comorbidity [Count of Participants; unit: Participants]
  Cardiovascular disease | 10 | 11 | 21
  Pulmonary disease | 3 | 3 | 6
  Diabetes mellitus | 0 | 4 | 4
  Previous breast cancer | 3 | 3 | 6
Current medication [Count of Participants; unit: Participants]
  Antidepressant/sedative | 2 | 3 | 5
  Analgesics | 5 | 2 | 7
ASA classification (American Society of Anesthesiologists physical status classification system) [Count of Participants; unit: Participants] — ASA Physical Status Classification (ASA I to VI) (ASA I: a normal healthy patient, ASA II: a patient with mild systemic disease, ASA III: a patient with severe systemic disease)
  Participants
    Class I | 9 | 11 | 20
    Class II | 15 | 13 | 28
    Class III | 1 | 1 | 2
EQ-5D health index preoperatively (EuroQol Group form five dimensions) [Median (Full Range); unit: score on a scale] — The EQ-5D is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 3-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Values are anchored at 1 (full health) and 0 (death) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead.
  score on a scale | 0.81 [0.12 to 1.00] | 0.82 [0.12 to 1.00] | 0.81 [0.12 to 1.00]
HADS Anxiety (Hospital Anxiety and Depression Scale) [Count of Participants; unit: Participants]
  No anxiety | 13 | 15 | 28
  Mild-moderate anxiety | 9 | 6 | 15
  Severe anxiety | 3 | 4 | 7
HADS Depression (Hospital Anxiety and Depression Scale) [Count of Participants; unit: Participants]
  No depression | 21 | 21 | 42
  Mild-moderate depression | 4 | 4 | 8
PSQ score (Pain Sensitivity Questionnaire score) [Median (Full Range); unit: score on a scale (0-10)] — The PSQ is composed of 17 items, describing a daily life situation, asking to rate pain on a scale from 0 (not painful) to 10 (worst pain). 3 of the 17 situations are not normally painful and not included in the PSQ-total score(=an average score;17-3=14 items/14). The PSQ-minor is calculated as the average of 7 items of mild pain intensity of 14 items. The PSQ-moderate score is the calculated average rating of 7 items of moderate pain intensity of 14 items. In all scores higher values represent a worse outcome. Range of all three scores min 0 to max 10.
  score on a scale (0-10)
    PSQ total score (range 0-10) | 2.9 [1.6 to 6.6] | 3.3 [0.4 to 6.6] | 3.1 [0.4 to 6.6]
    PSQ minor score (range 0-10) | 2.1 [0.6 to 5.0] | 2.3 [0.3 to 7.3] | 2.3 [0.3 to 7.3]
    PSQ moderate score(range 0-10) | 4.4 [1.0 to 9.7] | 4.4 [0.6 to 7.3] | 4.4 [0.6 to 9.7]

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life (HRQoL)
Description: Quality of life measured by means of the EuroQol form (EQ-5D). The EQ-5D form was completed daily during the first eight days after surgery, then once weekly for additional six weeks. The health state index has a possible range from 0 to 1 with a higher score meaning a better quality of life.
Time Frame: Days 0, 1, 2, 3, 4, 5, 6, 7, 14, 21, 28, 35, 42
Population: Women with low-risk early stage endometrial cancer scheduled for radical surgery at the University Hospital in Linköping between February 2012 and may 2016 were asked to participate int the study according to the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
scores on a scale
  EQ-5D Day 0 | 0.34 (0.40) | 0.30 (0.53)
  EQ-5D Day 1 | 0.66 (0.24) | 0.48 (0.40)
  EQ-5D Day 2 | 0.74 (0.19) | 0.56 (0.31)
  EQ-5D Day 3 | 0.73 (0.19) | 0.59 (0.28)
  EQ-5D Day 4 | 0.77 (0.19) | 0.63 (0.30)
  EQ-5D Day 5 | 0.83 (0.18) | 0.64 (0.31)
  EQ-5D Day 6 | 0.84 (0.17) | 0.67 (0.25)
  EQ-5D Day 7 | 0.83 (0.22) | 0.66 (0.29)
  EQ-5D Day 14 | 0.88 (0.11) | 0.73 (0.22)
  EQ-5D Day 21 | 0.91 (0.12) | 0.71 (0.31)
  EQ-5D Day 28 | 0.92 (0.10) | 0.76 (0.29)
  EQ-5D Day 35 | 0.93 (0.12) | 0.82 (0.26)
  EQ-5D Day 42 | 0.95 (0.09) | 0.86 (0.22)
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.011, ANOVA — Main effect over time p<0.001; Interaction effect p=0.65. Threshold for statistical significance p<0.05

2. Secondary Outcome: Changes in Biomarkers for Tissue Damage (C-reactive Protein (hsCRP))
Description: The biomarker was measured on seven occasions. Time 1: one week before surgery. Time 2: just before surgery. Time 3: two hours postoperatively. Time 4: 24 hours postoperatively. Time 5: 48 hours postoperatively. Time 6: one week after surgery. Time 7: six weeks after surgery.
Time Frame: One week and just before surgery. Two, 24 and 48 hours postoperatively. One and six weeks after surgery.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
mg/L
  hsCRP time 1 | 2.5 (2.1) | 6.0 (17.0)
  hsCRP time 2 | 2.7 (2.6) | 4.7 (11.4)
  hsCRP time 3 | 2.3 (2.3) | 3.5 (6.7)
  hsCRP time 4 | 29.0 (29.4) | 52.3 (27.0)
  hsCRP time 5 | 46.3 (49.8) | 75.4 (43.7)
  hsCRP time 6 | 10.5 (8.6) | 9.3 (8.6)
  hsCRP time 7 | 2.9 (2.6) | 1.9 (1.5)
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.03, ANOVA — P-value main effect between groups. Effect over time p < 0.0001. Interaction effect p 0.02. Threshold for statistical significance p<0.05; Tukey post hoc test (p-values): hsCRP time 4 p 0.02; hsCRP time 5 p <0.001

3. Secondary Outcome: Changes in Biomarkers for Tissue Damage (White Blood Cells (WBC))
Description: as for outcome 2
Time Frame: One week and just before surgery. Two, 24 and 48 hours postoperatively. One and six weeks after surgery.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: x10^9 cells/L
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
x10^9 cells/L
  WBC time 1 | 6.7 (1.7) | 7.7 (2.1)
  WBC time 2 | 6.2 (1.7) | 6.6 (1.7)
  WBC time 3 | 6.8 (3.0) | 11.4 (3.7)
  WBC time 4 | 9.4 (3.3) | 10.1 (2.8)
  WBC time 5 | 7.2 (2.3) | 9.2 (2.3)
  WBC time 6 | 7.2 (2.0) | 7.6 (2.0)
  WBC time 7 | 6.5 (1.5) | 6.8 (1.6)
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p < 0.01, ANOVA — P-value main effect between groups. Effect over time p < 0.0001. Interaction effect p < 0.0001. Threshold for statistical significance p < 0.05; Tukey post hoc test (p-value): WBC time 3 p < 0.0001

4. Secondary Outcome: Changes in Biomarkers for Tissue Damage (Interleukin 6 (IL-6))
Description: as for outcome 2
Time Frame: One week and just before surgery. Two, 24 and 48 hours postoperatively. One and six weeks after surgery.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
pg/ml
  IL-6 time 1 | 15.0 (29.8) | 10.9 (19.0)
  IL-6 time 2 | 15.7 (29.0) | 9.6 (13.8)
  IL-6 time 3 | 21.0 (28.7) | 47.6 (24.5)
  IL-6 time 4 | 28.0 (31.0) | 37.9 (19.0)
  IL-6 time 5 | 15.3 (21.8) | 17.3 (9.4)
  IL-6 time 6 | 18.4 (31.2) | 10.0 (12.1)
  IL-6 time 7 | 13.1 (25.7) | 12.2 (28.8)
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.03, ANOVA; Tukey post hoc test (p-value): IL-6 time 3 p < 0.01

5. Secondary Outcome: Changes in Biomarkers for Tissue Damage (Creatin Kinase (CK))
Description: as for outcome 2
Time Frame: One week and just before surgery. Two, 24 and 48 hours postoperatively. One and six weeks after surgery.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µkat/L
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
µkat/L
  CK time 1 | 1.8 (1.1) | 1.6 (1.1)
  CK time 2 | 1.9 (1.1) | 1.6 (1.0)
  CK time 3 | 1.5 (0.9) | 2.5 (1.0)
  CK time 4 | 3.3 (2.5) | 6.2 (4.9)
  CK time 5 | 3.0 (2.4) | 4.5 (2.1)
  CK time 6 | 1.0 (0.6) | 0.9 (0.6)
  CK time 7 | 1.6 (1.1) | 1.3 (0.8)
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.03, ANOVA — P-value main effect between groups. Effect over time p < 0.0001. Interaction effect p < 0.01. Threshold for statistical significance p < 0.05; Tukey post hoc test (p-value): CK time 4 p < 0.0001

6. Secondary Outcome: Changes in Biomarkers for Tissue Damage (Cortisol)
Description: as for outcome 2
Time Frame: One week and just before surgery. Two, 24 and 48 hours postoperatively. One and six weeks after surgery.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
nmol/L
  Cortisol time 1 | 273.4 (75.0) | 266.0 (123.2)
  Cortisol time 2 | 489.0 (137.0) | 510.1 (131.2)
  Cortisol time 3 | 301.0 (267.0) | 533.2 (249.0)
  Cortisol time 4 | 392.0 (201.0) | 383.0 (178.1)
  Cortisol time 5 | 358.1 (128.0) | 379.0 (125.4)
  Cortisol time 6 | 309.1 (98.0) | 331.0 (76.0)
  Cortisol time 7 | 307.0 (129.0) | 331.1 (125.4)
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.06, ANOVA — [p-value comment as in outcome 5, analysis 1]; Tukey post hoc test (p-value): cortisol time 3 p < 0.0001

7. Secondary Outcome: Health Economics (With 300 Robotic Procedures Annually)
Description: Total costs (direct and indirect) for hospital stay and recovery period until six weeks postoperatively.
Time Frame: From the day of surgery until six weeks after surgery.
Measure: Number; unit: Swedish crowns per procedure
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
Swedish crowns per procedure
  Direct costs per procedure | 65,728 | 46,776
  Indirect costs per procedure | 12,451 | 18,318
  Total costs (direct + indirect) per procedure | 78,179 | 65,094
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.06, t-test, 2 sided

8. Secondary Outcome: Health Economics (With 500 Robotic Procedures Annually)
Description: Total costs (direct and indirect) for hospital stay and recovery period until six weeks postoperatively.
Time Frame: From the day of surgery until six weeks after surgery.
Measure: Number; unit: Swedish crowns per procedure
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
Number analyzed (Participants) | 25 | 24
Swedish crowns per procedure
  Direct costs per procedure | 61,862 | 46,769
  Indirect costs per procedure | 12,451 | 18,318
  Total costs (direct + indirect) per procedure | 74,313 | 65,087
Statistical Analysis 1: Comparison: Robotic Hysterectomy vs Abdominal Hysterectomy; Test type: Superiority; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the day of surgery until six weeks postoperatively.
Arm/Group | Robotic Hysterectomy | Abdominal Hysterectomy
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 2/24
Other Adverse Events (participants affected / at risk) | 8/25 | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Hysterectomy (N=25) | Abdominal Hysterectomy (N=24)
Reoperation vaginal vault bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Hysterectomy (N=25) | Abdominal Hysterectomy (N=24)
Wound complications (Infections and infestations) | 0 (0) | 6 (6)
Neuralgia (Nervous system disorders) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vaginal vault hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Red blood cell transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spinal punction not possible (Surgical and medical procedures) | 1 (1) | 2 (2)
Intubation difficulties (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Nothing to declare.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No